CLINICAL TRIAL: NCT01658202
Title: Nicotine Patch Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: V00116 TD 1 04; 2011-006212-32 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-06 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Healthy Smokers
Keywords: Smoking cessation; Nicotine; Tobacco Use Disorder; Central Nervous System Agents
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

ARMS (2):
- Sequence 1 (Other): After a 24h washout period free of any nicotine exposure, subjects will be randomly assigned to one of 2 treatment-sequence groups, separated by a 48h-intervals.
  Each patch will be applied for 24h.
  Interventions: Drug: V0116 transdermal patch (Test treatment ); Drug: Nicotine transdermal patch (Reference Treatment )
- Sequence 2 (Other): After a 24h washout period free of any nicotine exposure, subjects will be randomly assigned to one of 2 treatment-sequence groups, separated by a 48h-intervals.
  Each patch will be applied for 24h.
  Interventions: Drug: V0116 transdermal patch (Test treatment ); Drug: Nicotine transdermal patch (Reference Treatment )

INTERVENTIONS:
Drug: V0116 transdermal patch (Test treatment )
Drug: Nicotine transdermal patch (Reference Treatment )

SUMMARY:
The purpose of this study is to compare the relative bioavailability of nicotine following single application of a new transdermal formulation to that of a reference formulation.

4 single 24hour applications separated by 48hour intervals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject aged 18 to 45 years (inclusive)
* Current Smoker of >or = 5 and < or = 15 cigarettes/day
* Fagerström score < or =5 at selection
* Absence of any clinically significant abnormal finding at physical, vital sign, Electrocardiogram ECG, biological examinations in the investigator's opinion.

Exclusion Criteria:

* Presence of any significant medical finding or significant history (in particular any cardio-vascular disease, severe renal or hepatic insufficiency, current gastric or duodenal ulcer) that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator
* Any visible skin disorder, abnormal skin pigmentation or dermatologic disease liable to interfere with use or assessment of transdermal patch

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | Blood samples will be collected on Days 1, 3, 5 and 7
  Pharmacokinetic profile of nicotine following a single patch application by measuring Maximum Plasma Concentration, Time of Maximum Concentration, Area under the nicotine plasma concentration curve, for each test and reference formulations

SECONDARY OUTCOMES:
Clinical safety (reported adverse events) | up to day 9
  General and local safety by evaluating the number of subjects with emergent adverse events or changes from baseline to end of study in vital signs, electrocardiogram, haematology and biochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes, France